CLINICAL TRIAL: NCT01726049
Title: Effects of Sildenafil on Pulmonary Arterial Pressure in Patients With Heart Failure With Preserved Ejection Fraction ( HFpEF) and Pulmonary Hypertension
Brief Title: Sildenafil in HFpEF (Heart Failure With Preserved Ejection Fraction) and PH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, E.S. Hoendermis, MD, PhD, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sildenafil Groningen Study
Record Dates: First submitted 2012-09-21; First posted 2012-11-14 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure, Diastolic; Pulmonary Hypertension
Keywords: HFpEF; PH
MeSH Terms: conditions — Heart Failure, Diastolic; Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil (Active Comparator): Sildenafil orally 3 times 20mg for 2 weeks , followed by 3 times 60 mg for 10 weeks
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): placebo orally 3 times 20mg tablets, followed by 3 times 60 mg for 10 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — Sildenafil administered orally 3 times per day 20 mg for the first 2 weeks, followed by 3 times 60 mg for 10 weeks
  Arms: Sildenafil
Drug: Placebo — Placebo tablets 3 times per day 20 mg foor de first 2 weeks, followed by 3 times 60 mg for 10 weeks
  Arms: Placebo

SUMMARY:
Aim of the study is to investigate whether Sildenafil treatment results in a reduction of pulmonary artery pressure without decrease of cardiac output (CO) and in improvement of exercise capacity in patients with heart failure with preserved ejection fraction (HFpEF) with pulmonary hypertension ( PH).

DETAILED DESCRIPTION:
Rationale: Treatment of diastolic left heart failure is a challenging task. Compared to systolic left heart failure the level of evidence for known medical treatment regiments is low. Sildenafil, a phosphodiesterase 5 (PDE 5) inhibitor and effective therapy for pulmonary arterial hypertension acts as a selective pulmonary vasodilator by inhibiting the impaired nitric oxide (NO) pathway. Reducing the pulmonary vascular resistance would be the primary target by treatment of diastolic left heart failure with PH. But clinical and hemodynamical studies to evaluate the role of Sildenafil in diastolic heart failure, also called heart failure with preserved ejection fraction (HFpEF) with secondary pulmonary hypertension are lacking. Our hypothesis is that Sildenafil decreases pulmonary artery pressure in patients with HFpEF and pulmonary hypertension.

Objective: To investigate whether Sildenafil treatment results in a hemodynamic improvement and in an improvement of exercise capacity in these patients.

Study design: single-center, prospective, randomized, placebo controlled study. Study population: 52 patients with HFpEF and PH Intervention : One group receives three times daily 20 mg Sildenafil for 2 weeks followed by three times daily 60 mg Sildenafil for 10 weeks. The other group receives three times daily 20 mg of Placebo, followed by 3 times daily 60 mg placebo.

Main study parameters/endpoints:

Primary objectives

1. To investigate whether Sildenafil treatment results in a reduction of pulmonary artery pressure (PAP) in HFpEF patients with PH (investigated invasively by right heart catheterization) .

Secondary objectives

1. To investigate whether Sildenafil treatment results in an reduction of wedge pressure in HFpEF patients.
2. To investigate whether Sildenafil treatment results in an improvenemt of cardiac output (CO) in HFpEF patients.
3. To investigate whether Sildenafil treatment results in improvement of exercise capacity in these patients ( defined as change in VO2max)

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Written inform consent
* PH secondary to diastolic left heart failure defined as
* PAP mean >25 mmHg
* Wedge mean >15 mmHg
* Normal systolic left ventricular (LV) function on echo/nuclear imaging (left ventricular ejection fraction (LVEF) > or =45%)
* New York Heart Association class (NYHA) II-IV despite heart failure therapy

Exclusion Criteria:

* Severe noncardiac limitation to exercise (as severe chronic obstructive pulmonary disease)
* Other cause of PH besides diastolic heart failure
* Coronary ischemia or recent myocardial infarction (<6 months)
* Hypotension ( <90/50 mmHg)
* Ongoing nitrate therapy
* Ongoing therapy with citochrome P450 3A4 ( CYP3A4) inhibitors (ketoconazole, erythromycin, cimetidine, clarithromycin, itraconazole, voriconazole and protease inhibitors) or CYP3A4 inductors(carbamacepine, phenytoin, phenobarbital, rifampicin, Sint Janskruid ). Furthermore patients will be informed not to drink grapefruit juice while on study medication because of the known impact of grape fruit on pharmacokinetics of Sildenafil.
* Ongoing therapy with alpha -inhibitors
* Significant mitral or aortic valve dysfunction
* Severe liver dysfunction
* Pregnancy
* Unable to read and comprehend Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-10; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E S Hoendermis, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Liu LC, Hummel YM, van der Meer P, Berger RM, Damman K, van Veldhuisen DJ, Voors AA, Hoendermis ES. Effects of sildenafil on cardiac structure and function, cardiopulmonary exercise testing and health-related quality of life measures in heart failure patients with preserved ejection fraction and pulmonary hypertension. Eur J Heart Fail. 2017 Jan;19(1):116-125. doi: 10.1002/ejhf.662. Epub 2016 Nov 21. PMID 27873388
- [Derived] Hoendermis ES, Liu LC, Hummel YM, van der Meer P, de Boer RA, Berger RM, van Veldhuisen DJ, Voors AA. Effects of sildenafil on invasive haemodynamics and exercise capacity in heart failure patients with preserved ejection fraction and pulmonary hypertension: a randomized controlled trial. Eur Heart J. 2015 Oct 7;36(38):2565-73. doi: 10.1093/eurheartj/ehv336. Epub 2015 Jul 17. PMID 26188003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Stabile outpatients with heart failure with preserved ejection fraction (HFpEF) and signs of pulmonary hypertension (PH) on echocardiogram were referred for right heart cath as part of clinical care. After heart catheter measurements , eligible patients were asked for participation. Recruitment from october 2011 until september 2014
Period: Overall Study
Arm/Group | Sildenafil | Placebo
Started | 26 | 26
Completed | 21 | 22
Not Completed | 5 | 4
Not completed — Death | 1 | 1
Not completed — Adverse Event | 4 | 1
Not completed — refused second HC | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil | Placebo | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (12) | 76 (7) | 74 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 6 | 9 | 15
Region of Enrollment [Number; unit: participants]
  Netherlands | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: Mean Pulmonary Artery Pressure Measured by Right Heart Catheterization
Description: change of mean pulmonary artery pressure between baseline and 12 weeks measured by heart catheterisation
Time Frame: baseline and 12 weeks
Population: 52 patients randomized. 26 Sildenafil arm: 26 placebo arm: change in mean pulmonary artery pressure could be evaluated in the intention to treat (ITT) analyses in 21 and 22 subjects of the Sildenafil and placebo treatment group
Measure: Mean (95% Confidence Interval); unit: mmHG
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 21 | 22
mmHG | -2.4 [-4.5 to -0.3] | -4.7 [-7.1 to -2.3]
Statistical Analysis 1: Comparison: Sildenafil; Test type: Superiority or Other; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-4.5 to -0.3]
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -4.7, 95% CI 2-sided [-7.1 to -2.3]

2. Secondary Outcome: VO2max
Description: difference in change of VO2 max between baseline and 12 weeks between Sildenafil and placebo group
Time Frame: baseline and 12 weeks
Population: 52 patients randomized. 26 Sildenafil arm: 26 placebo arm: change in VO2max could be evaluated in the ITT analyses in 18 and 22 subjects of the Sildenafil and placebo treatment group
Measure: Mean (95% Confidence Interval); unit: ml/kg/min
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 18 | 22
ml/kg/min | 0.2 [-0.9 to 1.4] | 0.7 [-0.3 to 1.6]
Statistical Analysis 1: Comparison: Sildenafil; Test type: Superiority or Other; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.9 to 1.4]
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-0.3 to 1.6]

3. Secondary Outcome: Cardiac Output Measured Invasively by Right Heart Catheterization
Description: difference in change of cardiac output between baseline and 12 weeks between Sildenafil and Placebo group
Time Frame: baseline and 12 weeks
Population: 52 patients randomized. 26 Sildenafil arm: 26 placebo arm: change in cardiac output could be evaluated in the ITT analyses in 20 and 22 subjects of the Sildenafil and placebo treatment group
Measure: Mean (95% Confidence Interval); unit: mililiter/min
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 20 | 22
mililiter/min | -0.4 [-0.9 to 0.1] | -0.2 [-0.5 to 0.1]
Statistical Analysis 1: Comparison: Sildenafil; Test type: Superiority or Other; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.9 to 0.1]
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.1]

4. Secondary Outcome: Wedge Pressure Measured Invasively by Right Heart Catheterization
Description: Difference in change of wedge pressure between baseline and 12 weeks between Sildenafil group and Placebo group
Time Frame: baseline and 12 weeks
Population: 52 patients randomized. 26 Sildenafil arm: 26 placebo arm: change in wedge pressure could be evaluated in the ITT analyses in 21 and 22 subjects of the Sildenafil and placebo treatment group
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 21 | 22
mmHg | -0.5 [-1.9 to 1.0] | -3.5 [-5.2 to -1.8]
Statistical Analysis 1: Comparison: Sildenafil; Test type: Superiority or Other; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.9 to 1.0]
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-5.2 to -1.8]

5. Other Pre Specified Outcome: Echocardiographic Parameters of Diastolic LV Dysfunction
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Sildenafil | Placebo
Serious Adverse Events (participants affected / at risk) | 4/26 | 3/26
Other Adverse Events (participants affected / at risk) | 22/26 | 21/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil (N=26) | Placebo (N=26)
intestinal infarction (Gastrointestinal disorders) | 0 | 1
cardiac failure (Cardiac disorders) | 1 | 0
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
pseudoaneurysma (Vascular disorders) | 1 | 0
medical device complication (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil (N=26) | Placebo (N=26)
headache (General disorders) | 4 | 3
nausea (Gastrointestinal disorders) | 2 | 2
dizziness (Nervous system disorders) | 1 | 3
visual impairment (Eye disorders) | 0 | 5
myalgia (Musculoskeletal and connective tissue disorders) | 4 | 4
respiratory tract infection (Infections and infestations) | 9 | 3
chest pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes